CLINICAL TRIAL: NCT02622789
Title: Efficacy and Influence of Pilates Based Physical Therapy Exercises on Spinal Radiographic Kinematics and Functional Status in Patients With Low Back Pain
Brief Title: Efficacy and Influence of Pilates Based Physical Therapy Exercises for Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: CRREC-104-081
Record Dates: First submitted 2015-11-08; First posted 2015-12-07 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Mechanical Low Back Pain
Keywords: Spinal alignment; Kinematics; Pilates; Physical Therapy
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Controls: Age-matched Healthy Controls
- General Exercises: Low Back Pain Participants Receiving General Exercises
- Pilates Exercises: Low Back Pain Participants Receiving Pilates Exercises
  Interventions: Other: Pilates Exercises

INTERVENTIONS:
Other: Pilates Exercises — Pilates method based stability exercise intervention
  Groups: Pilates Exercises

SUMMARY:
An assessment of the effectiveness of Pilates based physical therapy exercises for patients with low back pain (LBP) and its influence on spinal movement and patient reported functional disability.

DETAILED DESCRIPTION:
Low back pain (LBP) is becoming a major public health problem associated with enormous economic burden on the modern society. Despite conservative interventions such as Pilates back exercises are routinely prescribed in clinical practice, most studies to date have only assessed its efficacy based on subjective patient reported outcomes with limited objective data available to clearly demonstrate the benefit of Pilates exercise on spinal alignment and mobility. Furthermore, patient adherence has been well identified to be an obstacle for effective home exercise program and the most cost-effective strategy to improve patient compliance remain unknown. Current study therefore aims to fulfil this gap in our knowledge by assessing the change of spinal alignment and kinematics utilizing dynamic radiographs performed pre- and post- a 6-week Pilates based physical therapy exercise program compare to a more generic hospital based back care exercise program. Furthermore, the effectiveness of conducing weekly phone reminders for 6 weeks on improving short (6-month) and long (12-month) term functional outcomes and patient compliance will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Predominant LBP for a minimum of three consecutive months as diagnosed by a rehabilitation physician

Exclusion Criteria:

1. . Radicular neurological signs,
2. . Trauma induced LBP,
3. . Diagnosis of spinal deformity such as scoliosis or spondylolisthesis,
4. . Spinal infection or tumor,
5. . Rheumatologic conditions,
6. . Previous spinal surgery,
7. . History of hip or pelvic disorder that required treatment,
8. . Contradiction for radiographic exposure such as pregnancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is anticipated that 100 patients with clinical signs and symptoms of low back pain (LBP) for at least 3 months will be recruited. 25 age-matched healthy control will also be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic Spino-pelvic Alignment Parameters | 12-month
  Thoroaco-lumbo-pelvic dynamic radiographs taken for both maximum flexion and extension will be analysed to determine parameters such as 1. Pelvic incidence angle, 2. Pelvic tilt angle, 3. Sacral slope angle, 4. Lumbosacral angle, 5. Lumbar lordosis angle and 6.
Radiographic Lumbar Spine Segmental and Global Range of Motion | 12-month
  Thoroaco-lumbo-pelvic dynamic radiographs taken for both maximum flexion and extension will be analysed to determine the lumbar spine segmental and its contribution to the global range of motion

SECONDARY OUTCOMES:
Modified Oswestry Disability Index | 12-month
  Questionnaires to determine patients' self-reported pain and functional disabilities
Roland Morris Disability Questionnaire | 12-month
  Questionnaires to determine patients' self-reported pain and functional disabilities
Short Form-36 | 12-month
  Questionnaires to determine patients' self-reported pain and functional disabilities

CONTACTS AND LOCATIONS:
Overall Officials: Andy Chien, PhD, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan